CLINICAL TRIAL: NCT02335684
Title: Improving Functional Capacity in Heart Failure Patients Supported With Continuous-flow Left Ventricular Assist Devices. -Effects of Increased Pump Speed During Sustained Submaximal Exercise
Brief Title: Effects of Increased CF-LVAD Pump Speed During Sustained Submaximal Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: H-1-2013-103
Record Dates: First submitted 2014-01-20; First posted 2015-01-12 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Heart-assist devices; exercise capacity
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- CF-LVAD patients. (Experimental): Patients are compared with themselves during submaximal exercise testing with baseline pump speed vs. submaximal exercise testing with increased pump speed.
  Interventions: Other: CF-LVAD pump speed baseline.; Other: CF-LVAD pump speed increased.

INTERVENTIONS:
Other: CF-LVAD pump speed baseline. — Submaximal exercise test with baseline pump speed.
Other: CF-LVAD pump speed increased. — Submaximal exercise test with increased pump speed (+800RPM).

SUMMARY:
This randomized trial has been designed to study if it is possible to enhance work capacity during submaximal efforts in heart failure patients supported with continuous-flow left ventricular assist devices (CF-LVAD).

The hypothesis is that exercise tolerability during low to moderate workloads in CF-LVAD patients can be increased when pump speed is increased soon after the onset of exercise.

DETAILED DESCRIPTION:
To test the hypothesis described above the investigators will study submaximal exercise tests below anaerobic threshold in patients supported with CF-LVADs.Each patient will perform two tests- one with baseline CF-LVAD pump speed and the other with incrementally increased pump speed.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic and non-ischemic cardiomyopathy patients with CF-LVADs,signed informed consent.

Exclusion Criteria:

* Unstable patients, CF-LVAD implantation less than three months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Exercise time | Exercise time will be estimated only on the day of the study. No follow-up.
  Exercise will be performed on a upright ergometer bike with simultaneously breath-by-breath gaz analysis.

SECONDARY OUTCOMES:
Perceived exertion | Perceived exertion will be estimated during exercise on the ergometer bike on the day of the study.
  Rate of exertion will be estimated using the Borg Scale.

OTHER OUTCOMES:
Heart rate | Heart rate will be measures during exercise.
  Heart rate is measured by ECG monitoring.
Anaerobic threshold | Anaerobic threshold is measured during exercise on the study day.
  Anaerobic threshold is defined as respiratory exchange rate (RER) >1.

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University Hospital of Copenhagen; Rigshospitalet., Copenhagen Oe, Denmark